CLINICAL TRIAL: NCT01728636
Title: The Use of Tranexamic Acid to Reduce Perioperative Blood Loss During High Risk Spine Fusion Surgery
Acronym: TXA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Louanne Carabini, Assistant Professor of Anesthesiology & Neurological Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00066949
Record Dates: First submitted 2012-11-09; First posted 2012-11-20 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Curvature of Spine
MeSH Terms: conditions — Spinal Curvatures | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Experimental): Tranexamic acid 10mg/kg loading dose given pre-incision and 1mg/kg/hr infusion throughout intraoperative period
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Normal saline placebo loading dose 0.5ml/kg and infusion at 0.5ml/kg/hr throughout operative course
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — intravenous administration of bolus and infusion for duration of surgical procedure
  Other Names: Lysteda

SUMMARY:
The purpose of this study is to determine if tranexamic acid reduces perioperative blood loss and red blood cell transfusion during high risk spine surgery.

DETAILED DESCRIPTION:
There are conflicting studies in the literature reporting different efficacy outcomes for the use of antifibrinolytics in spine fusion surgery. Several studies support the successful use of tranexamic acid for major orthopedic procedures, but the patient populations studied for spine surgery thus far have been small and highly variable, with less than clinically significant results. If TXA if efficacious in reducing not only perioperative blood loss, but RBC transfusion without an increase in thromboembolic events, then its use may be justified for patients at risk for major blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* age>17 years
* undergoing posterior spine fusion surgery for kyphoscoliosis with a >80% chance of major transfusion

Exclusion Criteria:

* age < 18 years
* non-English speaking
* pregnancy
* emergency procedures
* surgery for tumor, trauma or infection
* severe coronary artery disease
* history of venous thromboembolism
* history of cerebral vascular accident
* history of renal insufficiency
* allergy to tranexamic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louanne M Carabini, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Elgafy H, Bransford RJ, McGuire RA, Dettori JR, Fischer D. Blood loss in major spine surgery: are there effective measures to decrease massive hemorrhage in major spine fusion surgery? Spine (Phila Pa 1976). 2010 Apr 20;35(9 Suppl):S47-56. doi: 10.1097/BRS.0b013e3181d833f6. PMID 20407351
- [Background] Yang BP, Ondra SL, Chen LA, Jung HS, Koski TR, Salehi SA. Clinical and radiographic outcomes of thoracic and lumbar pedicle subtraction osteotomy for fixed sagittal imbalance. J Neurosurg Spine. 2006 Jul;5(1):9-17. doi: 10.3171/spi.2006.5.1.9. PMID 16850951
- [Background] Bernard AC, Davenport DL, Chang PK, Vaughan TB, Zwischenberger JB. Intraoperative transfusion of 1 U to 2 U packed red blood cells is associated with increased 30-day mortality, surgical-site infection, pneumonia, and sepsis in general surgery patients. J Am Coll Surg. 2009 May;208(5):931-7, 937.e1-2; discussion 938-9. doi: 10.1016/j.jamcollsurg.2008.11.019. Epub 2009 Mar 26. PMID 19476865
- [Background] Ferraris VA, Davenport DL, Saha SP, Austin PC, Zwischenberger JB. Surgical outcomes and transfusion of minimal amounts of blood in the operating room. Arch Surg. 2012 Jan;147(1):49-55. doi: 10.1001/archsurg.2011.790. PMID 22250113
- [Background] Henry D, Carless P, Fergusson D, Laupacis A. The safety of aprotinin and lysine-derived antifibrinolytic drugs in cardiac surgery: a meta-analysis. CMAJ. 2009 Jan 20;180(2):183-93. doi: 10.1503/cmaj.081109. Epub 2008 Dec 2. PMID 19050037
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, McClelland B, Laupacis A, Fergusson D. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD001886. doi: 10.1002/14651858.CD001886.pub2. PMID 17943760
- [Background] Kagoma YK, Crowther MA, Douketis J, Bhandari M, Eikelboom J, Lim W. Use of antifibrinolytic therapy to reduce transfusion in patients undergoing orthopedic surgery: a systematic review of randomized trials. Thromb Res. 2009 Mar;123(5):687-96. doi: 10.1016/j.thromres.2008.09.015. Epub 2008 Nov 12. PMID 19007970
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Elwatidy S, Jamjoom Z, Elgamal E, Zakaria A, Turkistani A, El-Dawlatly A. Efficacy and safety of prophylactic large dose of tranexamic acid in spine surgery: a prospective, randomized, double-blind, placebo-controlled study. Spine (Phila Pa 1976). 2008 Nov 15;33(24):2577-80. doi: 10.1097/BRS.0b013e318188b9c5. PMID 19011538
- [Background] Endres S, Heinz M, Wilke A. Efficacy of tranexamic acid in reducing blood loss in posterior lumbar spine surgery for degenerative spinal stenosis with instability: a retrospective case control study. BMC Surg. 2011 Nov 3;11:29. doi: 10.1186/1471-2482-11-29. PMID 22047046
- [Background] Gill JB, Chin Y, Levin A, Feng D. The use of antifibrinolytic agents in spine surgery. A meta-analysis. J Bone Joint Surg Am. 2008 Nov;90(11):2399-407. doi: 10.2106/JBJS.G.01179. PMID 18978408
- [Background] Tsutsumimoto T, Shimogata M, Ohta H, Yui M, Yoda I, Misawa H. Tranexamic acid reduces perioperative blood loss in cervical laminoplasty: a prospective randomized study. Spine (Phila Pa 1976). 2011 Nov 1;36(23):1913-8. doi: 10.1097/BRS.0b013e3181fb3a42. PMID 21289587
- [Background] Halpin RJ, Sugrue PA, Gould RW, Kallas PG, Schafer MF, Ondra SL, Koski TR. Standardizing care for high-risk patients in spine surgery: the Northwestern high-risk spine protocol. Spine (Phila Pa 1976). 2010 Dec 1;35(25):2232-8. doi: 10.1097/BRS.0b013e3181e8abb0. PMID 21102298
- [Background] Tzortzopoulou A, Cepeda MS, Schumann R, Carr DB. Antifibrinolytic agents for reducing blood loss in scoliosis surgery in children. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD006883. doi: 10.1002/14651858.CD006883.pub2. PMID 18646174
- [Background] Dirkmann D, Gorlinger K, Gisbertz C, Dusse F, Peters J. Factor XIII and tranexamic acid but not recombinant factor VIIa attenuate tissue plasminogen activator-induced hyperfibrinolysis in human whole blood. Anesth Analg. 2012 Jun;114(6):1182-8. doi: 10.1213/ANE.0b013e31823b6683. Epub 2011 Nov 21. PMID 22104068
- [Background] Ozier Y, Bellamy L. Pharmacological agents: antifibrinolytics and desmopressin. Best Pract Res Clin Anaesthesiol. 2010 Mar;24(1):107-19. doi: 10.1016/j.bpa.2009.09.014. PMID 20402174

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 31 | 30
Completed | 31 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Median (Full Range); unit: Years] | 68 [62 to 72] | 65 [62 to 69] | 66 [62 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61
Weight (kilogram) [Mean (Standard Deviation); unit: kilogram (kg)] — Weight measured in kilograms
  kilogram (kg) | 82.1 (18.9) | 72.9 (21.7) | 77 (20)
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 165.9 (9.4) | 161.7 (11.6) | 163 (11)
Body Mass Index [Mean (Full Range); unit: kg/m^2] — Body mass index calculated by: kg/m^2
  kg/m^2 | 31.2 [24.3 to 33.8] | 26.4 [22.7 to 30.8] | 29 [22.7 to 33.8]
ASA status [Mean (Full Range); unit: score on a scale] — American Society of Anesthesiologists Physical Status.
  1. Healthy person.
  2. Mild systemic disease.
  3. Severe systemic disease.
  4. Severe systemic disease that is a constant threat to life.
  5. A moribund person who is not expected to survive without the operation.
  6. A declared brain-dead person whose organs are being removed for donor purposes.
  score on a scale | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]
Medical History (none) [Count of Participants; unit: Participants] — No contributory medical history.
  Participants | 6 | 12 | 18
History of hypertension [Count of Participants; unit: Participants] | 13 | 21 | 34
History of coronary artery disease [Count of Participants; unit: Participants] | 0 | 2 | 2
History of atrial fibrillation [Count of Participants; unit: Participants] | 1 | 0 | 1
History of peripheral vascular disease [Count of Participants; unit: Participants] | 1 | 0 | 1
History of diabetes melitus [Count of Participants; unit: Participants] | 3 | 7 | 10
History of asthma [Count of Participants; unit: Participants] | 3 | 3 | 6
History of obstructive sleep apnea [Count of Participants; unit: Participants] | 4 | 4 | 8
Baseline Hemoglobin (g/dl) [Mean (Standard Deviation); unit: g/dl (grams per deciliter)] — Hemoglobin measured as grams per deciliter/
  g/dl (grams per deciliter) | 10.6 (1.0) | 10.6 (1.4) | 10.6 (1.2)
Baseline hematocrit [Mean (Standard Deviation); unit: Percent] — Baseline hematocrit in %.
  Percent | 32.1 (2.9) | 31.9 (4) | 32 (3.4)
Baseline Platelets [Mean (Inter-Quartile Range); unit: x 10^5 cells/mm^3] — Baseline platelets x 10^5 cells/mm^3
  x 10^5 cells/mm^3 | 136 [120 to 149] | 133 [112 to 146] | 135 [112 to 149]
Baseline fibrinogen (mg/dL) [Mean (Full Range); unit: miligrams per deciliter] — Fibrinogen measured in miligrams per deciliter.
  miligrams per deciliter | 272 [222 to 321] | 268.5 [239 to 347] | 270 [222 to 347]
Preoperative risk of major transfusion [Mean (Full Range); unit: Percent] — The preoperative risk of receiving a major blood transfusion described as percent risk.
  0%= no preoperative risk- 100% high risk. Above 100%-600% very high risk.
  Percent | 212 [130 to 505] | 505 [150 to 550] | 358 [130 to 550]
Total number of vertebral levels [Mean (Full Range); unit: Vertebra levels] — Total number of vertebral levels operated upon.
  Vertebra levels | 15 [10 to 16] | 10 [9 to 16] | 13 [9 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Total Red Blood Cells Transfused in the Intraoperative Period
Description: Total red blood cells transfused in the intraoperative period in (mL). Total RBC equal packed red blood cells and cell saver infusion.
Time Frame: Intraoperative period (approximately 12 hours)
Measure: Median (Inter-Quartile Range); unit: milliliters
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 31 | 30
milliliters | 1140 [560 to 1744] | 1460 [1115 to 2650]
Statistical Analysis 1: Comparison: Tranexamic Acid vs Placebo; Test type: Superiority; p = .05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Additional Blood Products Transfused
Description: Total additional blood products (fresh frozen plasma, cryoprecipitate, and platelets) transfused in the perioperative period measured in units.
Time Frame: 24 hours after skin incision
Measure: Mean (Full Range); unit: Units
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 31 | 30
Units | 1 [1 to 4] | 2 [0 to 4]

3. Secondary Outcome: Post Operative Major Morbidity
Description: Number of participants who experienced arterial or venous thromboembolism, neurologic complications (including stroke, seizure,and delirium), infections, and pulmonary renal or cardiac adverse outcomes (demand ischemia, myocardial infarction or new arrhythmia) before another operative procedure or hospital discharge.
Time Frame: Time of surgery to date of discharge from hospital (average 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 31 | 30
Participants | 9 | 9

4. Other Pre Specified Outcome: Estimated Intraoperative Blood Loss
Description: Estimated Intraoperative blood loss in milliliters (mLs)
Time Frame: Incision to skin closure (approximately 10 hours)
Measure: Mean (95% Confidence Interval); unit: Milliliters
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 31 | 30
Milliliters | 1550 [1200 to 3200] | 1600 [1200 to 2500]

5. Other Pre Specified Outcome: Total Tranexamic Acid Dose (mg)
Description: Total milligrams of intravenous tranexamic acid administered during the surgical procedure.
Time Frame: Intraoperative period
Measure: Median (Full Range); unit: milligrams
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 31 | 30
milligrams | 1408 [1235 to 1685] | 0 [0 to 0]

6. Post Hoc Outcome: Total Operating Room Time
Description: Total operating room time from incision to closure of incision in minutes.
Time Frame: Minutes
Measure: Median (Full Range); unit: Minutes
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 31 | 30
Minutes | 602 [522 to 653] | 576 [526 to 690]

ADVERSE EVENTS:
Time Frame: Start of surgery to discharge from the hospital ( approximately 7 days)
Arm/Group | Tranexamic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 9/31 | 9/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=31) | Placebo (N=30)
Composite outcome of postoperative adverse events (General disorders) | 9 (9) | 9 (9) — The events cannot be separated. Data was reported as composite outcome of postoperative morbidity including arterial or venous thromboembolic , renal or neurologic morbitity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT01728636/Prot_SAP_000.pdf